CLINICAL TRIAL: NCT01880632
Title: A Multicenter, Single Arm, Open-label Trial of Oxaliplatin Plus Capecitabine (XELOX) in the Perioperative Treatment of Locally Advanced Gastric Adenocarcinoma
Brief Title: Oxaliplatin Plus Capecitabine in the Perioperative Treatment of Locally Advanced Gastric Adenocarcinoma
Acronym: Neo-Classic
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Ruijin Hospital (Other); RenJi Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Tianshu Liu, Director of Medical oncology derpartment, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28733
Record Dates: First submitted 2013-06-08; First posted 2013-06-19 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Gastric Adenocarcinoma
Keywords: XELOX; perioperative treatment; locally advanced gastric adenocarcinoma; D2 resection
MeSH Terms: interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- XELOX (Experimental): Clinically diagnosed stage T2-3/N+M0,orT4aN+M0 according to CT/MRI scan, and resectable
  Interventions: Drug: XELOX

INTERVENTIONS:
Drug: XELOX — Patients will be given the perioperative chemotherapy as below once recruited:
  Capecitabine ：500 mg tablets（Roche） Oxaliplatin：50mg/10ml（according to daily practice in each center）
  Schedule of Oxaliplatin plus capecitabine (XELOX) will be as follow:
  Capecitabine 1000 mg/m2 ，orally taken 30 minutes after meal, bid ， d 1~14 every 3 weeks(treatment for 2 weeks and rest 1 week) Oxaliplatin：130mg/m2， iv infusion over 2h，d1,every 3 weeks

SUMMARY:
1. Target population:locally advanced gastric adenocarcinoma (LAGC, cT2~3/N+M0,or cT4aN+M0);no previous chemo or radio therapy.
2. Primary objective:Response rate of XELOX in the neoadjuvant setting of LAGC.

   Secondary objectives:
   * The progression free survival (PFS) in the perioperative treatment of locally advanced gastric adenocarcinoma (cT3/N+M0,or cT4aN+M0);
   * percentage of pathological response ; percentage of grade 3 or 4 adverse events as safety profile of perioperative treatments;
   * D2 resection -rate after neoadjuvant chemotherapy of XELOX;
   * Overall survival;
   * QOL during the whole period of treatment.
3. Trial design:This is a multicenter, single arm, open-label, phase II study to evaluate the efficacy and safety of Oxaliplatin plus capecitabine(XELOX) in the perioperative treatment of locally advanced gastric adenocarcinoma in combination with D2 resection.
4. Treatment plan:Patients will be given the perioperative chemotherapy as below once recruited:Schedule of Oxaliplatin plus capecitabine (XELOX) will be as follow: Capecitabine 1000 mg/m2 ，bid,d 1~14 every 3 weeks(treatment for 2 weeks and rest 1 week)Oxaliplatin：130mg/m2， iv infusion over 2h，d1,every 3 weeks.
5. Number of subjects:50 patients.Number of centers 5 sites, which have the high volume of gastric operations in China, more than 500 per year.

DETAILED DESCRIPTION:
1. Disease specific inclusion criteria:

   * Histologically documented gastricadenocarcinoma with Lauren classification Clinically diagnosed stage T2-3/N+M0,orT4aN+M0 according to CT/MRI scan, and resectable
   * Measurable disease is required
   * Karnofsky score 80%.
   * Physical condition and adequate organ function to ensure the success of abdominal surgery.
   * Life expectancy ≥12 weeks.
   * Adequate hematological function: Neutrophil count ≥ 1.5 × 109/L, Platelets ≥ 100 × 109/L and Hemoglobin ≥8g/dL .Adequate liver function: Total bilirubin ≤ 1.5 × upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) < 2.5 × ULN in the absence of liver metastases, or < 5 × ULN in case of liver metastases. ALP ≤ 2.5 × upper limit of normal (ULN); ALB ≥30g/L.

   Adequate renal function: Serum creatinine ≤ 1.25 x ULN, and creatinine clearance ≥ 60 ml/min.
   * Female subjects should not be pregnant or breast-feeding.
   * No serious concomitant disease that will threaten the survival of patients to less than 5 years.
2. General inclusion criteria:

   * Male or female. Age ≥ 18 years and ≤75 years
   * Written (signed) informed consent.
   * Able to comply with study and follow-up procedures.
   * Good compliance with the treatment plan。
   * Consent to provide tissue sample。

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented gastricadenocarcinoma with Lauren classification Clinically diagnosed stage T2-3/N+M0,orT4aN+M0 according to CT/MRI scan, and resectable
* Measurable disease is required
* Karnofsky score 80%.
* Physical condition and adequate organ function to ensure the success of abdominal surgery.
* Life expectancy ≥12 weeks.
* Adequate hematological function: Neutrophil count ≥ 1.5 × 109/L, Platelets ≥ 100 × 109/L and Hemoglobin ≥8g/dL .Adequate liver function: Total bilirubin ≤ 1.5 × upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) < 2.5 × ULN in the absence of liver metastases, or < 5 × ULN in case of liver metastases. ALP ≤ 2.5 × upper limit of normal (ULN); ALB ≥30g/L.Adequate renal function: Serum creatinine ≤ 1.25 x ULN, and creatinine clearance ≥ 60 ml/min.
* Female subjects should not be pregnant or breast-feeding.
* No serious concomitant disease that will threaten the survival of patients to less than 5 years.
* Male or female.
* Age ≥ 18 years and ≤75 years
* Written (signed) informed consent.
* Able to comply with study and follow-up procedures.
* Good compliance with the treatment plan.
* Consent to provide tissue sample.

Exclusion Criteria:

* Pregnant or lactating (in case of potentially childbearing woman, pregnancy test is positive)
* Patients of child-bearing age or the potential to father a child who refuse to use adequate contraception
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* History of another malignancy in the last 5 years with the exception of the following:

Any previous palliative, adjuvant or neoadjuvant chemotherapy and/or radiotherapy. Prior treatment for locally advanced or metastatic gastric cancer. Any metastatic disease will render patient ineligible according to AJCC staging manual.

* Distant metastases (M1) including distant nodal Groups (peripancreatic, para-aortic, portal, retroperitoneal, mesenteric node, by CT/MRI, or PET/CT
* Treatment within the last 30 days with any investigational drug. Concurrent administration of any other cancer therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Poorly controlled diabetes mellitus with fasting blood sugar > 18 mM. Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* History of significant neurological or mental disorder, including seizures or dementia, which would interfere compliance and sign of consent inform. any history of hypersensitivity to 5-fluorouracil or platinum and other investigational drug
* Ileus, chronic inflammatory intestinal disease or extensive resection of the small intestine and other disorders which limit drug reabsorption. This includes gastric dumping syndrome, indications of accelerated passage through the small intestine, indications of reabsorption disorders after intestinal surgery
* Unstable, persistent cardiac disease despite medicinal treatment, myocardial infarction within 6 months before the start of the trial
* Organ transplant patient need immunosuppression treatment.
* Previous surgery on primary tumour; Prior palliative surgery (open and closure, passage operation)
* Any other type of tumour (e.g. leiomyosarcoma, lymphoma) or a secondary malignancy, excepting basal cell skin carcinoma or basal cell carcinoma in situ of the cervix which have already been successfully treated
* Symptomatic peripheral neuropathy NCI CTC version> 3.0 grade.
* Patients under anticoagulant therapy with warfarin or other coumarines are excluded from participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-05 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
the response rate of XELOX in the neoadjuvant setting of LAGC | 6 months after the last subject participating in
  the response rate evaluation will be based on tumor assessment with follow-up, including chest and upper-abdominal During preoperative treatment period, CT scan will be performed every 6 -8 weeks (2 cycles after)., brain MRI and bone scan (ECT) will be performed if any suspected symptoms occur.

SECONDARY OUTCOMES:
the progression free survival (PFS) in the perioperative treatment of locally advanced gastric adenocarcinoma (cT2-3/N+M0,or cT4aN+M0) | 42 months after the last subject participating in
  progression by the evidence of CT/MRI scan at each evaluation at neoadjuvant period or follow-up time after surgery；During preoperative treatment period, CT scan will be performed every 6 -8 weeks (2 cycles after).After syrgery, CT scan will be planned every 6 months, brain MRI and bone scan (ECT) will be performed if any suspected symptoms occur.
percentage of pathological response | 10 months after the last subject participating in
  After surgery，the pathological response will be measured by the pathologist for every Operation patient.
Percentage of grade 3 or 4 adverse events as safety profile of perioperative treatments | 1 month after the last date of treatment
  Adverse events and clinical laboratory tests will be recorded by CTCAE (version 4.0) during the whole treatment period.
Overall survival | 3 years after the last subject participating in
  During the OS follow-up, out-patient clinic and telephone visit will be done every 3 months for the first two years, and every 6 months after two years.
QOL during the whole period of treatment | 1 years after the last date of treatment
  These assessment will be evaluated at every evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu Liu, Doctor, Principal Investigator — Medical oncology Shanghai zhongshan hospital
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yu Y, Fang Y, Shen Z, Wang Y, Yan M, Cao H, Liu Y, Wang X, Cui Y, Liu F, Chen W, Li W, Li Q, Jiang H, Sun Y, Liu T. Oxaliplatin plus Capecitabine in the Perioperative Treatment of Locally Advanced Gastric Adenocarcinoma in Combination with D2 Gastrectomy: NEO-CLASSIC Study. Oncologist. 2019 Oct;24(10):1311-e989. doi: 10.1634/theoncologist.2019-0416. Epub 2019 Jun 25. PMID 31239311